CLINICAL TRIAL: NCT05386641
Title: Risk Factors for Shoulder Joint Motion Restriction in Breast Cancer Survivors
Brief Title: Risk Factors for Shoulder Joint Motion Restriction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Nilufer Kablan, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: 2022/0226
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer Survivors
Keywords: breast cancer; range of motion
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Breast cancer survivors with shoulder joint motion restriction
  Interventions: Other: measurement of tissue stiffness (N/m); Other: measurement of passive muscle tone (Hz); Other: measurement of creep of tissue; Other: measurement of the range of shoulder joint motion; Other: measurement of skin temperature; Other: measurement of pain; Other: measurement of pain pressure threshold; Other: measurement of grip strength
- Control group: Breast cancer survivors without shoulder joint motion restriction
  Interventions: Other: measurement of tissue stiffness (N/m); Other: measurement of passive muscle tone (Hz); Other: measurement of creep of tissue; Other: measurement of the range of shoulder joint motion; Other: measurement of skin temperature; Other: measurement of pain; Other: measurement of pain pressure threshold; Other: measurement of grip strength

INTERVENTIONS:
Other: measurement of tissue stiffness (N/m) — Stiffness values will be measured with myotonPro on centers of coordination located along the myofascial chain
Other: measurement of passive muscle tone (Hz) — muscle tones will be measured with myotonPro on centers of coordination located along along the myofascial chain
Other: measurement of creep of tissue — creep of tissue will be measured with myotonPro on centers of coordination located along the myofascial chain
Other: measurement of the range of shoulder joint motion — The range of shoulder flexion, abduction, extension and external-internal rotation movements will be measured with a universal goniometer.
Other: measurement of skin temperature — measurements will be taken by the thermographic camera
Other: measurement of pain — Pain will be evaluated by visual analog scale (VAS)
Other: measurement of pain pressure threshold — Pain pressure threshold will be evaluated by a digital algometer
Other: measurement of grip strength — The grip strength of both hand will be evaluated by "hand-held" dynamometer.

SUMMARY:
In breast cancer patients, limitation of shoulder joint movement may occur following cancer treatment. Shoulder limitation causes a significant decrease in the patient's participation in activities of daily living. The aim of the study is to define these limitations, to evaluate in detail all the structures that cause the problem, and to determine the causes of the limitations in patients with shoulder joint movement limitation developed after breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 30-60
* Having breast cancer treatment within 5 years

Exclusion Criteria:

* Not having agreed to participate in the study
* Presence of additional orthopedic (scoliosis, etc.), neurological (multiple sclerosis, stroke, etc.) and rheumatological diseases (ankylosing spondylitis, rheumatoid arthritis, etc.) that will affect upper extremity functions

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — breast cancer survivors
Study Population: Breast cancer survivors with or without shoulder joint restriction will be evaluated
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
measurement of tissue stiffness (N/m) | Baseline
  Stiffness values will be measured with myotonPro on centers of coordination located along the myofascial chain
measurement of passive muscle tone (Hz) | Baseline
  muscle tones will be measured with myotonPro on centers of coordination located along the myofascial chain
measurement of creep of tissue | Baseline
  creep of tissue will be measured with myotonPro on centers of coordination located along the myofascial chain
measurement of the range of shoulder joint motion | Baseline
  The range of shoulder flexion, abduction, extension and external-internal rotation movements will be measured with a universal goniometer.

SECONDARY OUTCOMES:
measurement of skin temperature | Baseline
  measurements will be taken from the area covering 3 cm of the surgical incision with a P45 thermographic camera with high thermal sensitivity
measurement of pain | Baseline
  Pain will be evaluated by visual analog scale (VAS). In the scale, the patient is asked to mark the most appropriate pain intensity on a scale ranging from 0 (no pain) to 10 (tolerable pain). The higher the score, the greater the pain intensity.
measurement of pain pressure threshold | Baseline
  Pain pressure threshold will be evaluated by a digital algometer
measurement of grip strength | Baseline
  The grip strength of both hand will be evaluated by "hand-held" dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University, Istanbul, Turkey (Türkiye)

REFERENCES:
- Available data/document: Individual Participant Data Set: 18192154 — https://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 25977305 — https://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 26079868 — http://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 29332760 — http://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 32031629 — http://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set: 32767329 — http://pubmed.ncbi.nlm.nih.gov/
- Available data/document: Individual Participant Data Set — http://pubmed.ncbi.nlm.nih.gov/